CLINICAL TRIAL: NCT04167293
Title: Effect of Stereotactic Body Radiotherapy Followed by Sintilimab Versus Stereotactic Body Radiotherapy Alone for Hepatocellular Carcinoma With Portal Vein Invasion After Arterially Directed Therapy: A Randomized Clinical Trial
Brief Title: Combination of Sintilimab and Stereotactic Body Radiotherapy in Hepatocellular Carcinoma (ISBRT01)
Acronym: ISBRT01
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mian XI (Other)
Responsible Party: Sponsor-Investigator, Mian XI, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-108-01
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; immunotherapy; PD-1; stereotactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT + PD-1 Arm (Experimental): Patients assigned to this arm will receive SBRT followed by sintilimab. Patients will receive stereotactic body radiotherapy (SBRT) using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3-6 fractions over 1-2 weeks. In the SBRT + PD-1 arm, sintilimab is administered intravenously at 200 mg every 3 weeks for up to 1 year. The first course of sintilimab will be given within 4-6 weeks after completion of SBRT.
  Interventions: Radiation: stereotactic body radiotherapy; Drug: Sintilimab
- SBRT Arm (Other): Patients assigned to this arm will receive SBRT alone. Patients will receive stereotactic body radiotherapy (SBRT) using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3-6 fractions over 1-2 weeks.
  Interventions: Radiation: stereotactic body radiotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — Patients will receive stereotactic body radiotherapy (SBRT) using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3-6 fractions over 1-2 weeks.
  Other Names: SBRT
Drug: Sintilimab — Sintilimab is administered intravenously at 200 mg every 3 weeks for up to 1 year. The first course of sintilimab will be given within 4-6 weeks after completion of SBRT.
  Other Names: IBI308
  Arms: SBRT + PD-1 Arm

SUMMARY:
Although sorafenib is the standard treatment for hepatocellular carcinoma with portal vein invasion, the outcome of these patients remains very poor, with a median survival time of 5.5 to 7.2 months. It has been demonstrated that first-line treatment with transarterial chemoembolization plus radiotherapy could provide more favorable survival than sorafenib alone. However, intrahepatic dissemination and distant metastasis remains the major recurrence pattern after treatment in these patients; therefore, searching for new strategies to improve efficacy is necessary. Immunotherapy targeting the PD-1/PD-L1 checkpoints has demonstrated promising activity in advanced HCC. Combining radiotherapy with immune checkpoints showed promising response rates and improved survival in several solid tumor types. The aim of this randomized study was to investigate the efficacy and safety of stereotactic body radiotherapy followed by sintilimab (an anti-PD-1 antibody) compared with stereotactic body radiotherapy alone for hepatocellular carcinoma with portal vein invasion after arterially directed therapy.

DETAILED DESCRIPTION:
A total of 116 HCC patients with portal vein invasion after arterially directed therapy (transarterial chemoembolization or hepatic arterial infusion chemotherapy) will be randomized to two treatment arms using a 1:1 ratio: SBRT + PD-1 arm or SBRT alone arm. Patients in both arms will receive stereotactic body radiotherapy (SBRT) using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3-6 fractions over 1-2 weeks. In the SBRT + PD-1 arm, sintilimab is administered intravenously at 200 mg every 3 weeks for up to 1 year. The first course of sintilimab will be given within 4-6 weeks after completion of SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed hepatocellular carcinoma or diagnosed by American Association for the Study of Liver Disease criteria;
2. No previous treatment for hepatocellular carcinoma, and received arterially directed therapy (transarterial chemoembolization or hepatic arterial infusion chemotherapy) as initial treatment and achieved technical success;
3. Absence of extrahepatic metastasis disease;
4. Portal vein invasion (at least the first- or second-branch portal vein) confirmed by 2 imaging techniques;
5. Less than 3 active intrahepatic lesions with a total diameter of less than 15 cm were required, at least one of which is measurable according to the mRECIST Criteria;
6. Age at diagnosis 18 to 75 years;
7. Eastern Cooperative Oncology Group performance status ≤ 2
8. Child-Pugh class A liver function;
9. Normal liver volume greater than 700 ml;
10. Estimated life expectancy ≥12 weeks;
11. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 3.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 50×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
12. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with systemic anti-tumor therapy (including chemotherapy, molecule-targeted therapy, immunotherapy, etc.);
2. Patients with extrahepatic metastasis disease at diagnosis;
3. The total diameter of the active intrahepatic lesions was more than 15 cm;
4. A history of abdominal radiotherapy;
5. Known or suspected allergy or hypersensitivity to monoclonal antibodies;
6. Patients who have a preexisting or coexisting bleeding disorder;
7. Female patients who are pregnant or lactating;
8. Inability to provide informed consent due to psychological, familial, social and other factors;
9. A history of malignancies other than hepatocellular carcinoma before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer;
10. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
11. Patients who cannot tolerate radiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia;
12. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
13. A history of interstitial lung disease or non-infectious pneumonia;
14. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
15. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay);
16. Any unstable situation that may endanger the safety and compliance of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2019-11-16 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
24-week progression-free survival (PFS) rate | 24 weeks after radiotherapy
  The proportion of patients with progression disease according to mRECIST at 24 weeks from randomization.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years from randomization
  From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
Overall survival (OS) | 2 years from randomization
  From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 24 months.
24-week overall response rate (ORR) | 24 weeks after radiotherapy
  The proportion of patients with complete response or partial response according to mRECIST at 24 weeks from randomization.
24-week disease control rate (DCR) | 24 weeks after radiotherapy
  The proportion of patients with complete response, partial response or stable disease according to mRECIST at 24 weeks from randomization.
Duration of response (DOR) | 2 years from randomization
  From date of first CR/PR to the date of first PD according to RECIST criteria, assessed up to 24 months.
Adverse Events | 2 years from randomization
  Treatment-related adverse events are graded according to the Common Toxicity Criteria, version 4.0, and were registered from the date of informed consent until discontinuation of trial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shi Y, Su H, Song Y, Jiang W, Sun X, Qian W, Zhang W, Gao Y, Jin Z, Zhou J, Jin C, Zou L, Qiu L, Li W, Yang J, Hou M, Zeng S, Zhang Q, Hu J, Zhou H, Xiong Y, Liu P. Safety and activity of sintilimab in patients with relapsed or refractory classical Hodgkin lymphoma (ORIENT-1): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2019 Jan;6(1):e12-e19. doi: 10.1016/S2352-3026(18)30192-3. PMID 30612710
- [Result] Shen L, Xi M, Zhao L, Zhang X, Wang X, Huang Z, Chen Q, Zhang T, Shen J, Liu M, Huang J. Combination Therapy after TACE for Hepatocellular Carcinoma with Macroscopic Vascular Invasion: Stereotactic Body Radiotherapy versus Sorafenib. Cancers (Basel). 2018 Dec 14;10(12):516. doi: 10.3390/cancers10120516. PMID 30558224
- [Result] Yoon SM, Ryoo BY, Lee SJ, Kim JH, Shin JH, An JH, Lee HC, Lim YS. Efficacy and Safety of Transarterial Chemoembolization Plus External Beam Radiotherapy vs Sorafenib in Hepatocellular Carcinoma With Macroscopic Vascular Invasion: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):661-669. doi: 10.1001/jamaoncol.2017.5847. PMID 29543938